CLINICAL TRIAL: NCT07350083
Title: Promoting Parental and Child Mental Health Through Emotion-focused Parenting Programs: Adaptation, Implementation, and Evaluation of Tuning in to Kids® in Portugal
Brief Title: Tuning in to Kids® for Parents of Preschool-aged Children in Portugal
Acronym: TIK-PT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lusofona University (Other)
Collaborators: Santa Casa da Misericórdia de Lisboa (Unknown); Aventura Social (Unknown); NucliSol Jean Piaget (Unknown); Pressley Ridge (Unknown); Associação Nacional de Apoio ao Desenvolvimento, Investigação e Comunidade (Unknown); Instituto Belong - Desenvolvimento e Saúde (Unknown); Associação de Aldeias de Crianças SOS (Unknown); Associação Passo a Passo (Unknown); CPCJ da Amadora (Unknown); CPCJ de Lisboa Ocidental (Unknown); Instituto de Apoio à Criança (Unknown); MSV - Crescer Como Família (Unknown); Unidade Local de Saúde Amadora-Sintra (Unknown); Comissão Nacional de Promoção dos Direitos e Proteção das Crianças e Jovens (Unknown); FUNDAÇAO CALOUSTE GULBENKIAN (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Stephanie Alves, Professor, Lusofona University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TIK-PT/FCG/335706; FCG/Growing Minds/335706 (Other Grant/Funding Number: Fundação Calouste Gulbenkian); UID/05380/2025 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2025-12-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Parental Emotion Socialization; Parents' Beliefs About and Reactions to Children's Emotions; Parental Emotion Regulation
Keywords: Tuning in to Kids®; parental emotion socialization; randomized controlled trial; preschool; children emotional and behavioral difficulties

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuning in to Kids® intervention (Experimental): Participants will attend a 6-week, in-person group program structured around emotion coaching principles (Tuning in to Kids®).
  Interventions: Behavioral: Tuning in to Kids®
- Waiting list group (Other): Participants will be offered and receive TIK after the conclusion of the final follow-up assessment.
  Interventions: Behavioral: Tuning in to Kids®

INTERVENTIONS:
Behavioral: Tuning in to Kids® — Tuning in to Kids® (TIK) is a manualized program delivered by trained facilitators (6 weekly - 2h - group sessions) and aimed to promote parents' emotion socialization practices that are supportive of the child's expression of emotion (emotion coaching; e.g., comforting, teaching constructive means of coping), while reducing unsupportive ESPP (emotion dismissing; e.g., punishing or minimizing). An additional booster session may be held after two months of program's conclusion. TIK includes strategies informed by emotion coaching principles, including psychoeducation, roleplays, video materials, mindfulness-based exercises, and group discussions. By addressing a core mechanism leading to different emotional and behavioral childhood disorders (i.e. difficulties in emotion regulation), TIK is susceptible to promoting children's long-term full potential and parental mental health outcomes.

SUMMARY:
Early parent-child interactions, namely how parents respond to their children's emotions (i.e., emotion socialization parenting practices [ESPP]), may play a critical role in how children develop emotion regulation abilities. When parents rely on unsupportive ESPP, this can result in regulatory problems, which are a transdiagnostic symptom of MH problems, being a major cause of its etiology. Emotion-focused parenting programs, such as Tuning in to Kids® (TIK), promote parents' emotion coaching skills, enabling children to understand and regulate their emotions in more effective ways, while also supporting parents in managing their own emotions.

This study aims to examine the feasibility, acceptability, implementation fidelity and efficacy of the TIK program among parents of preschool-aged children in Portugal. TIK is a 6-week group, face-to-face program grounded in the principles of emotion coaching, among other theoretical backgrounds such as Mindfulness and Emotion Regulation Theories.

This trial is a parallel two-arm randomized clinical trial. Participants will be parents/legal guardians (> 18 years old) with at least one child between 3 and 6 years old and with proficiency in portuguese. At least 152 parents/legal guardians will be recruited with the support of several community partners. Interested parents will be contacted by telephone to confirm their eligibility. Participants will be informed about their eligibility during the intake interview, followed by a full explanation of the clinical trial procedures. Eligible participants will be randomly assigned to either the intervention group (TIK) or a waitlist control group, with the latter receiving the intervention after the follow-up assessment. The intervention consists of six weekly in-person group sessions plus one follow-up session, each lasting approximately 2 hours. Participants in both groups will complete questionnaires at three time points - baseline, post-intervention, and 2-month follow-up - covering different dimensions of children (e.g., children's emotional and developmental difficulties) and parental (e.g., parenting stress) psychological functioning, and parenting (e.g., ESPP).

ELIGIBILITY:
Inclusion Criteria:

Parents/legal guardians:

* with at least one child aged between 3 and 6 years old (inclusive) who lives with the parent/legal guardian,
* with at least 18 years old,
* who can read, understand, and speak Portuguese
* who live in the Lisbon Metropolitan Area or Lisbon District. When applicable, both parents will be allowed to participate.

Exclusion Criteria:

* parents' poor Portuguese language skills
* parents' being currently enrolled in another structured parenting program
* if the target child is already attending elementary school at the time of recruitment
* if the target child has a diagnosis of a severe Communication and/or Developmental Disorder, or
* if the target child is under a child protection measure that implies that the child does not live with their parents (e.g., if the child is in foster care).

Only participants that give informed consent to participate in the study will be included and randomized to one of the study conditions (TIK vs. waiting list group).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in parents' beliefs about children's emotions | Baseline, immediately post-intervention, and 2 months follow-up
  Measured with the Parents' Beliefs About Children's Emotions Questionnaire (PBACE). The PBACE is a 33-item self-report questionnaire, with items rated on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). The present study will use the following subscales: Value of Anger, Manipulation, Control, and Autonomy. Subscale scores will be calculated by averaging item responses, with higher scores indicating stronger endorsement of the corresponding belief in that category.
Changes from baseline in parents' reactions to children's emotions | Baseline, immediately post-intervention, and 2 months follow-up
  Measured with the Coping with Children's Negative Emotions Scale (CCNES). The CCNES is a parent-report measure assessing how parents respond to children's negative emotions across 12 hypothetical scenarios, with responses rated on a 7-point Likert scale from 1 (very unlikely) to 7 (very likely). The CCNES comprises seven subscales: Emotion-Focused, Problem-Focused, Expressive Encouragement, Minimizing, Punitive, Distress, and Ignoring reactions. Items from the first three subscales are summed to create a composite measure of emotion coaching, whereas items from the remaining four subscales are summed to assess emotion dismissing responses. For each scale, total scores are calculated by averaging item responses, with higher scores indicating greater endorsement of the corresponding practice.
Changes from baseline in parents' emotion regulation (parenting-specific) | Baseline, immediately post-intervention, and 2 months follow-up
  Measured with the Interpersonal Mindfulness in Parenting Scale (IM-P). The IM-P is a 29-item self-report instrument rated on a 5-point Likert scale, from 1 (never true) to 5 (always true). The Self-Regulation in Parenting will be assessed as primary outcome. Subscale scores will be calculated by summing item responses. Higher scores on the Self-Regulation in Parenting subscale indicate greater ability to regulate emotions and behaviors within the parenting context.
Changes from baseline in parents' emotional regulation (general) | Baseline, immediately post-intervention, and 2 month follow-up
  Measured with the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF). The DERS-SF is a self-report measure, including 18 items, rated on a 5-point Likert scale, ranging from 1 (almost never) to 5 (almost always). A total score is obtained by averaging all items, with higher scores indicating greater difficulties. In line with the recommendations of the Portuguese authors, items 1, 4 and 6 will be excluded from the analyses.

SECONDARY OUTCOMES:
Changes from baseline in children's behavioral and emotional difficulties | Baseline, immediately post-intervention, and 2 month follow-up
  Measured with the Strengths and Difficulties Questionnaire - Parent (SDQ-P). The SDQ-P is a self-report measure for parents, including 25 items, each rated on a 3-point Likert scale, from 0 (not true) to 2 (certainly true). The total difficulties score is calculated by summing the scores from the following subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, and Peer Relationship Problems. Higher scores reflect greater difficulties. The Prosocial Behavior subscale is scored separately, as a measure of strengths. Two age-specific versions will be presented to parents (for children aged 3-4 and 5-6). The versions differ slightly in wording, but share the same scoring method and interpretation.
Changes from baseline in children' emotional regulation | Baseline, immediately post-intervention, and 2 month follow-up
  Measured with the Emotion Regulation Checklist (ERC). The ERC is a self-report measure consisting of 20 items rated on a 4-point Likert scale, ranging from 1 (never) to 4 (almost always). The ERC comprises two subscales: Emotion Regulation, and Emotion Lability/Negativity. For each subscale, a total score is obtained by the sum of the items. Higher scores on the Emotion Regulation subscale indicate higher emotion regulation; whereas higher scores on the Lability/Negativity subscale indicate higher difficulties in emotion regulation.
Changes from baseline in parenting stress | Baseline, immediately post-intervention, and 2 month follow-up
  Measured with the Parental Stress Scale (PSS). The PSS is a self-report scale comprising 18 items rated on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree). A total score is calculated by summing all items, with higher scores reflecting higher levels of parenting stress. Following the recommendations from the Portuguese authors, items 1-2 and 17-18 will be excluded from the analyses.
Changes from baseline in depressive symptoms | Baseline, immediately post-intervention, and 2 month follow-up
  Measured with the Depressive Symptoms subscale of the Hospital Anxiety and Depression Scale (HADS). This subscale consists of 7 items rated on a 4-point Likert scale, from 0 to 3 (e.g., "not at all", "most of the time"). The total score is obtained by summing the scores of the items, with higher scores being indicative of higher levels of depressive symptoms.
Changes from baseline in parenting self-efficacy | Baseline, immediately post-intervention, and 2 month follow-up
  Measured with the Self-Efficacy subscale of the Me as a Parent Questionnaire (MaaP). This subscale consists of 4 items rated on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree). A total score is obtained by adding up the items, with higher scores reflecting higher levels of perceived self-efficacy.

OTHER OUTCOMES:
Acceptability of the intervention | Immediately post-intervention
  Measured using a 16-item Likert-scale questionnaire developed by the research team; scores ranging from 1 (not at all) to 5 (very much). The questionnaire evaluates: (1) overall satisfaction with TIK; (2) the extent to which TIK met parents' expectations and contributed to improvements in parents' self-confidence, parent-child relationships, children's well-being, and parents' ability to understand and manage their children's emotions; (3) the frequency of applying TIK strategies in daily interactions; (4) the adequacy of the number, length and frequency of sessions; (5) satisfaction with the group format; (6) perceptions of facilitator competence and the intervention facilities; and (7) the perceived long-term usefulness of the acquired strategies. Participants will also indicate whether they would recommend the program to other parents (yes/no) and rate the ease of understanding and applying emotion coaching strategies on a scale from 1 (very easy) to 5 (very difficult)
Feasibility of the intervention | Immediately post-intervention
  Measured by participant adherence to the sessions, and facilitators and barriers to implementation. Adherence is measured by session attendance, with completion defined as attending at least 4 out of 6 sessions (i.e., 67%). Participants missing sessions will be contacted to identify barriers to participation. Regardless of completion, all participants will report factors that helped or hindered participation. Dropouts will be contacted to determine specific reasons, and the timing of dropout will be recorded. Overall attrition will be measured by the number of participants not completing post-intervention and/or follow-up assessments.
Implementation fidelity of the intervention | During the intervention (at the end of each session).
  Both facilitators and an independent observer (present in all groups) will complete the TIK Program Fidelity Checklist. For each planned activity outlined in the intervention manual, they will indicate whether the content was delivered as intended, with space provided for additional comments or notes.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology and Life Sciences, Lusófona University, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
Collective results from this trial will be shared to scientific and non-scientific communities after its conclusion.